CLINICAL TRIAL: NCT01895491
Title: An Open-Label, Uncontrolled, Single Center, Phase I Trial to Assess the Safety of VM206RY in Subjects With Expression of Her2 in Breast Cancer
Brief Title: Safety Study of VM206RY in Subjects With Expression of HER2 in Breast Cancer
Acronym: VM206RY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reyon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VM206RY-VM01
Record Dates: First submitted 2013-06-12; First posted 2013-07-10 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CohortⅠ (Experimental): VM206DNA 6mg and VM206Ad 3*10^9VP injected into the brachial muscle
  Interventions: Biological: VM206DNA; Biological: VM206Ad
- CohortⅡ (Experimental): VM206DNA 12mg and VM206Ad 3*10^9VP injected into the brachial muscle
  Interventions: Biological: VM206DNA; Biological: VM206Ad
- CohortⅢ (Experimental): VM206DNA 24mg and VM206Ad 3*10^9VP injected into the brachial muscle
  Interventions: Biological: VM206DNA; Biological: VM206Ad

INTERVENTIONS:
Biological: VM206DNA
Biological: VM206Ad

SUMMARY:
The main objective of this study is to evaluate the safety of VM206RY in subjects with expression of HER2 in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women, 20 years of age
* Stage 3 or 4 breast cancer
* Unresectable breast cancer with Expression of Her2 and one of the following criteria including

  * Prior use of Her2-targeted therapies(Herceptin, Tykerb, taxane and capecitabine) but it was not responding, with Immunohistochemistry (IHC) 3+, or IHC 2+ and FISH+, or SISH+
  * Patients received treatment that three times continuously Different chemotherapies but it was not responding, with Immunohistochemistry (IHC) 2+ and FISH- or SISH-, or Immunohistochemistry (IHC) 1+
  * Prior use of six chemotherapies(Anthracycline, Taxane, Gemcitabine, Capecitabine, Vinorelbine, Cyclophosphamide) but it was not responding, with Immunohistochemistry (IHC) 2+ and FISH or SISH-, or Immunohistochemistry (IHC) 1+
* One or more measurable(or assessable) lesion of breast or metastatic site

  * Spiral CT: ≥ 10mm diameter
  * general measurement methods (CT, X-ray, MRI): ≥ 20mm diameter
* Life expectancy 6 months
* Signed informed consent

Exclusion Criteria:

* Prior use of breast cancer vaccine
* Active or history of cardiovascular diseases within the past 3 months: Active uncontrolled cardiac disease, including cardiomyopathy, CHF(NYHA Class III~IV), and unstable angina, family history of congenital long QT syndrome or QT/QTc interval >0.45 sec or torsade de points(TdP), and history of idiopathic ventricular tachycardia or ventricular fibrillation, LVEF < 50%
* Patients with coronary artery disease (myocardial infarction, angina, etc.) or a history of coronary artery disease
* Patients who is required hospitalization by severe fever or required antibiotic treatment by serious infection
* Patients who is confirmed as CNS metastases. (Only, patient with stable brain metastases is permit. Among the patients who have not any symptom, do not see the progression before registered the last 2 month)
* History of prior malignancies other than breast cancer within the past 5 years
* Patients with an existing condition or a history of autoimmune disease or immunodeficiency disease
* ECOG score ≥ 3
* Patients with severe dysfunction in major organs

  * Blood: WBC < 3,000/㎕; Platelet < 100,000/㎕; Hematocrit < 30
  * Liver: Total bilirubin ≥ 1.5 x ULN; ALT/AST ≥ 2.5 x ULN
  * Kidney: Creatinine ≥ 1.5 x ULN
* Abnormal values of anti-nuclear Ab, anti-double-stranded DNA and C3, as judged by the investigator
* History of surgical procedure, chemotherapy, Herceptin treatment, corticosteroid therapy, immunosuppressant therapy or radiotherapy within the past 4 weeks
* HIV Ag/Ab, HBs Ag, HCV Ab or HTLV-1 Ab positive
* Psychotropic drug misuse/abuse or alcoholism
* Prior use of vaccine within the past 4 weeks
* Cumulative dose of prior doxorubicin > 360 ㎎/㎡ or epirubicin > 720 ㎎/㎡
* Women who is pregnant or breastfeeding and don't agree to use a contraceptive during the study period.
* Patients who have participated in clinical trials enrolled in this clinical trial within 4 weeks before. (Only patient, who has taken survey and DNA test without drug-treatment, has permit.)
* Patients who are ineligible to participate in this study, as judged by the investigator.
* Patients who prohibit administering GM-CSF and prior use of GM-CSF within the past 4 weeks.
* Patients who expect hypersensitivity to investigational product (VM206RY) or any component of product.
* Due to malignancy neoplasm, patients who require supplementary oxygen or has severe dyspnea at rest
* Patients with hypertension [inadequately controlled hypertension (systolic > 180 mm Hg or diastolic > 100 mm Hg)] or a history of hypertension

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Adverse events (including serious adverse events and adverse events lead to treatment discontinuation) will be described according to severity and to their relationship with the study drug and injection procedure. | Up to 24 weeks

SECONDARY OUTCOMES:
Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD) | Up to 8 weeks
  DLT was defined as adverse events higher than grade 3 based on NCI CTCAE version 4.0 with respect to their relationship with the study drug and injection procedure until 2 weeks after final injection. MTD was defined as the highest dose evaluated for which less than 1/3 of the participants experienced DLT.
Analysis of HER2 specific antibody formation in plasma at pre and post injection using ELISA or FACS | Up to 24 weeks
Analysis of HER2 specific CTL response on PBMC at pre and post injection using IFN-gamma ELISPOT | Up to 24 weeks
Assessment of tumor response based on the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) | Up to 24 weeks
Change of HER2 level in plasma at pre and post injection using ELISA | Up to 24 weeks
Analysis of GM-CSF level in plasma at pre and post injection using ELISA | Up to be confirmed as negative
Analysis of VM206Ad in whole blood at pre and post injection using Q-PCR | Up to be confirmed as negative

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea